CLINICAL TRIAL: NCT03005496
Title: The Effect of Zinc, Beta-carotene, and Vitamin D3 Supplementation as Pro-inflammation Mediated Regulator in Preterm Delivery Through Placental Protein Adaptor MyD88 and TRIF, Transcription Factor NFkB, and Pro-inflammatory Cytokine IL-1β
Brief Title: The Effect of Zinc, β-carotene, and Vitamin D3 in Preterm Delivery Through Placental MyD88, TRIF, NFkB, and IL-1β
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rima Irwinda, MD, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 50/UN.2F1/ETIK/2016
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: PreTerm Birth
MeSH Terms: conditions — Premature Birth | interventions — Zinc; picolinic acid; Nifedipine; beta Carotene; Cholecalciferol; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Placebo Comparator): * Nifedipin 4x10 mg oral
  * Dexamethasone 2x6 mg iv for 2 days
  * Zinc 50 mg/day
  * Beta-carotene 25,000 IU
  * Vitamin D3 50,000 IU/weekly
  Interventions: Drug: Zinc; Drug: Nifedipine; Drug: Beta Carotene; Drug: Vitamin D3; Drug: Dexamethasone
- Control (Active Comparator): * Nifedipin 4x10 mg
  * Dexamethasone 2x6 mg iv for 2 days
  Interventions: Drug: Nifedipine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Zinc — included in intervention arm
  Other Names: Zinc Picolinate 50 mg
  Arms: Intervention
Drug: Nifedipine — included in intervention and control arm
  Other Names: Nifedipine 10 mg
Drug: Beta Carotene — included in intervention arm
  Other Names: Beta carotene 25,000 IU
  Arms: Intervention
Drug: Vitamin D3 — included in intervention arm
  Other Names: Cholecalciferol 50,000 IU
  Arms: Intervention
Drug: Dexamethasone — included in intervention and control arm
  Other Names: Dexamethasone 6 mg

SUMMARY:
This study is a controlled trial which compares the effect of zinc, beta-carotene, and Vitamin D3 supplementation in pregnant women which has preterm birth. The measured outcome is zinc, vitamin A, and 25(OH)D level in serum and placenta, MyD88, TRIF, NFκB, and IL-1β levels in placenta.

DETAILED DESCRIPTION:
The research will be held in Cipto Mangunkusumo General and Budi Kemuliaan Hospital.

Each participant of each group will be given the medication of preterm birth hospital protocol, which includes nifedipine 4x10 mg as tocolytic agent, dexamethasone 2x6 mg intravenous for 2 days which aims to support lung maturation, and antibiotic. Then, the blood sample is obtained for zinc, vitamin A and 25(OH)D levels examination. Subjects will be divided into 2 groups which are group whose given the oral zinc 50 mg/day, oral beta-carotene 25,000 IU and oral vitamin D3 50,000 IU/week supplementation, and group who is not given the intervention. Each participant will be observed until delivery. After delivery, level of zinc, vitamin A, and 25(OH)D in serum and placenta will be measured, as well as level of MyD88, TRIF, NFκB, and IL-1β in placenta.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who has preterm birth in 26-36 weeks gestational age

Exclusion Criteria:

* Multiple pregnancy
* Drug allergy
* Intra Uterine Growth Retardation (IUGR) is detected
* Congenital malformation in fetus was found
* Preterm Premature Rupture of Membrane (PPROM)
* Maternal complication such as gestational hypertension, preeclampsia, gestational diabetes mellitus, heart disease, infection, and autoimmune disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
placenta MyD88 | 1 year
  Placenta MyD88 will be measured by immunochemistry. The level will be compared between intervention and control group (percentage)
placenta TRIF | 1 year
  Placenta TRIF will be measured by immunochemistry. The level will be compared between intervention and control group (percentage)
Placenta NFkB | 1 year
  Placenta NFkB will be measured by immunochemistry. The level will be compared between intervention and control group (percentage)
Placenta 25(OH)D | 1 year
  Placenta 25(OH)D will be measured by LC-MS. The level will be compared between intervention and control group (ng/mL)
Placenta vitamin A | 1 year
  Placenta vitamin A will be measured by LC-MS. The level will be compared between intervention and control group (ng/mL)
Placenta zinc | 1 year
  Placenta zinc will be measured by ICP-MS. The level will be compared between intervention and control group (ug/L)
Placenta IL-1B | 1 year
  Placenta IL-1B will be measured by ELISA. The level will be compared between intervention and control group (pg/mL)
Serum zinc | 1 year
  Serum zinc will be measured by ICP-MS. The level will be compared between intervention and control group (ug/L)
Serum 25(OH)D | 1 year
  Serum 25(OH)D will be measured by LC-MS. The level will be compared between intervention and control group (ng/mL)
Serum vitamin A | 1 year
  Serum vitamin A will be measured by LC-MS. The level will be compared between intervention and control group (ng/mL)

IPD SHARING:
Plan to Share IPD: Yes
The research findings will be disseminated via publication of results, submission of information to public accessible databases, or meetings